CLINICAL TRIAL: NCT01423903
Title: Phase 1, Open-label, Multiple Dose Escalation Trial to Determine Safety and Tolerability of Once-Daily OPB-51602 in Subjects With Advanced Cancer
Brief Title: Phase 1, Open-label Trial to Determine Safety of OPB-51602 in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 266-09-202
Record Dates: First submitted 2011-08-03; First posted 2011-08-26 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Cancer
Keywords: Phase I; STAT-3 inhibitor; solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPDC-51602 (Experimental): Subjects with advanced solid tumors will be treated with OPDC-51602 once daily by mouth
  Interventions: Drug: OPB-51602

INTERVENTIONS:
Drug: OPB-51602 — A cycle will consist of 28 days of OPB-51602 be taken by study subjects daily by mouth for every day of each 28 day cycle.

SUMMARY:
The purpose of this study is to determine whether OPB-51602 is safe and tolerable when given daily by mouth to subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is based on data that support a role for the signal transducer and activator of transcription (STAT) family of proteins in oncogenesis. One of the mechanisms of action of OPB-51602 includes inhibition of STAT3 phosphorylation. Therefore OPB-51602 is expected to be active as an anti-cancer drug. This first-in-human study will characterize the safety profile of OPB-51602, evaluate the pharmacokinetics of OPB-51602, identify a recommended phase II dose, and obtain preliminary efficacy data, in subjects with advanced cancers for whom there is no standard treatment available.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years
2. Pathologically confirmed advanced cancer that is resistant or refractory to standard therapy or for which no standard curative therapy is available
3. At least 4 weeks since the last dose of prior chemotherapy, radiation therapy, or investigational agent.
4. Subjects must have recovered from adverse effects of prior therapy at time of enrollment to ≤ Grade 1 (excluding alopecia)
5. ECOG performance status ≤ 1
6. Life expectancy of ≥ 3 months following study entry
7. Adequate organ function, defined as follows:

   * Serum creatinine < 1.5 x the upper limit of normal (ULN)
   * Aspartate aminotransferase and alanine aminotransferase levels ≤ 3.0 x ULN (≤ 5.0 x ULN in the presence of known liver metastasis)
   * Total bilirubin ≤ 1.5 x ULN
   * Alkaline phosphatase levels ≤ 2.5 x ULN (≤ 5 x ULN in presence of bone metastasis)
   * Absolute neutrophil count of ≥ 1,500/mm³ (≥ 1.5 x 10⁹/L)
   * Platelet count ≥ 100,000/mm³ (≥ 100 x10⁹/L)
   * Hemoglobin ≥ 9 g/dL
8. For women of childbearing potential (WOCBP), a negative serum pregnancy test result at screening and negative urine pregnancy test on Day 1
9. WOCBP or men whose sexual partners are WOCBP must agree to use 2 methods of adequate contraception
10. Before any protocol-specific screening procedures are performed, subjects must have signed and dated the IRB-approved ICF.

Exclusion Criteria:

1. Uncontrolled concurrent illness, including ongoing or active infection, uncontrolled hypertension,or any other condition that could raise the subject's safety risk.
2. Altered mental status, psychiatric illness, or social situation that could limit compliance with study requirements and/or confound interpretation of study results.
3. Known infection with human immunodeficiency virus, hepatitis B, or hepatitis C.
4. Known brain metastasis that has not been treated and stable for at least 4 weeks, or subjects with leptomeningeal disease.
5. Subjects unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with absorption of oral drugs.
6. A history of major surgery within 28 days of first receipt of study drug. Subjects must have recovered fully from any surgery.
7. Nursing or pregnant women
8. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in opinion of investigator, contraindicates use of an investigational drug, or that may render subject at excessively high risk for treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of OPB-51602 | Weekly for first cycle, then every 2 weeks (on average up to 8 weeks).
  AEs, vital signs, body weight, ECGs, clinical laboratory tests, and performance status will be assessed.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OPB-51602 and to determine the MTD of OPB-51602 | 28 days
  The following PK parameters (Cmax, tmax, AUC₀-t, AUCtau, CLss/F and t½,z) will be determined using a non-compartmental approach for OPB-51602 and selected metabolites after single (Cycle 1, Day 1) and multiple daily doses (Cycle 2, Day 1).
Pharmacodynamic profile: | 28 days
  Study drug effects on STAT-3 phosphorylation will be assessed in PBMCs of study subjects in the dose escalation and expansion stages.
Antitumor effects: | Every 2 cycles (on average 8 weeks).
  Treatment response and/or disease progression in subjects with measurable disease will be evaluated after every 2 cycles using Response Evaluation Criteria in Solid Tumors (RECIST₉).

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Elekes, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (3):
- United States (3):
  - Sarasota, Florida
  - Boston, Massachusetts
  - Nashville, Tennessee